CLINICAL TRIAL: NCT05500430
Title: Clinical Evaluation of Bioactive Injectable Hybrid Resin Composite Restoration With or Without Air Abrasion Surface Pretreatment in the Repairing Capacity of Defective Composite Restoration, A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Air Abrasion Surface Pretreatment in the Repairing Capacity of Defective Composite Restoration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Salah Abdel-Aty hassan, Assistant lecturer, conservative department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: repair defective restoration
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Repair
Keywords: repair; defective restoration; sandblasting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surface pretreatment sandblasting (Experimental): Air abrasion sandblasting aluminum oxide particles (Al2O3) Aqua Care single (London, UK) will be done for the defective area then repairing with bioactive injectable composite, Beautiful Flow Plus X F00 (Shofu, Japan).
  The surface treatment for aged composite will be applied according to manufacturer instructions.
  Repairing with bioactive injectable composite, Beautiful Flow Plus X F00(Shofu, Japan) The material will be applied according to manufacturer instructions. After shade selection incremental insertion in layers not exceeding 2 mm and light curing for 10 sec using 3M Eliper curing unite (Elipar Deepcure-S, 3M).
  Interventions: Device: Air abrasion sandblasting aluminum oxide particles (Al2O3) AquaCare single (Velopex, Medivance Instruments Ltd., London, UK)
- Repairing with conventional nanohybrid composite (Active Comparator): The nanohybrid resin composite will be applied to the the cavity using the conventional incremental technique according to manufacturer instructions.
  Interventions: Device: Air abrasion sandblasting aluminum oxide particles (Al2O3) AquaCare single (Velopex, Medivance Instruments Ltd., London, UK)

INTERVENTIONS:
Device: Air abrasion sandblasting aluminum oxide particles (Al2O3) AquaCare single (Velopex, Medivance Instruments Ltd., London, UK) — Air abrasion sandblasting aluminum oxide particles (Al2O3) Aqua Care single (London, UK) will be done for the defective area then repairing with bioactive injectable composite, Beautiful Flow Plus X F00 (Shofu, Japan).
  Other Names: sandblasting

SUMMARY:
This study is conducted to compare the efficacy of surface pretreatment using air abrasion sandblasting aluminum oxide particles (Al2O3) versus not pretreatment in the repair capacity of defective composite restoration indicated for repair.

DETAILED DESCRIPTION:
First the rationale for the repair, rather than the replacement of defective direct composite restorations proved a less invasive procedure with decreased tooth loss avoiding weakening and overtreatment of tooth. Less traumatic or stressful than replacement for patients with good acceptance; Increased longevity of the restoration; Reduction of potentially harmful effects on the dental pulp and Less risk of iatrogenic damage to adjacent teeth.

Secondary using surface treatment strategies aim to prepare a clean surface with high surface energy to provide better wettability with adequate surface roughness and surface area by removing the superficial layer of the aged composite which lead to increase integrity between old and new resin restoration.

ELIGIBILITY:
Inclusion Criteria:

* Co-operative patients approving to participate in the trial.
* patient with occlusal defects class I or class II composite resin restorations indicated for repair.

Exclusion Criteria:

* Allergic history concerning methacrylate.
* Rampant caries.

  * Disabilities patient
  * Pregnancy
  * Heavy smoking.
  * Xerostomia.
  * Lack of compliance.
  * Evidence of parafunctional habits.
  * Temporomandibular joint disorders.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in the clinical performance | Change from the baseline at 12 months
  Change in the clinical performance Measured using modified USPHS criteria for clinical evaluation of restoration failure.
  Measuring Unit:
  Scoring system (Ordinal):
  * Alfa
  * Bravo
  * Charlie
  * Delta

CONTACTS AND LOCATIONS:
Overall Officials: heba hamza, Professor, Study Director — heba.hamza@dentistry.cu.edu.eg
Locations (1):
- Dentistry, Cairo, Egypt